CLINICAL TRIAL: NCT06528795
Title: The Effect of Hybrid Simulation-Based Lactation Consultancy Training on Midwifery Students' Psychosocial Care Competence and Communication Skills
Brief Title: The Effect of Hybrid Simulation-Based Lactation Consultancy Training on the Skills of Midwifery Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBÜ-AYDINKARTAL-006
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Breastfeeding Consultancy Training
Keywords: Hybrid Simulation; Midwifery Students; Psychosocial Care Competence; Communication Skill

STUDY DESIGN:
Intervention Model Description: Quasi-experimental randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (n:40) (Experimental): Intervention group students will be practiced with the "Lactation Simulator", a high-reality simulator, in the simulation laboratory, accompanied by a scenario.
  Lactation Simulation Model (LSM) is a high fidelity simulator and is an applied and wearable breastfeeding model that educators can use for interactive training. LSM can be worn like a t-shirt and is placed over the shoulders and placed on the chest, then secured with a seat belt from the back. Thus, the seat belt can be adjusted for every size and weight. LSM is a simulator with the ability to respond to hand manipulation.
  Thanks to this feature, simulated milk release occurs when pressure is applied to the breast tissue, which is approximately 3 cm behind both nipples. It is also a suitable model for expressing milk by hand or with a pump. LSM has four different skin tones. The fact that LSM can be applied on clothing contributes significantly to the protection of privacy.
  Interventions: Other: Scenario-based high-reality hybrid simulation method
- Control group (n:40) (No Intervention): Control group students will practice on a simple breast model within the scope of classical education.
  Simple Breast Model: Can be used to teach and practice breast palpation techniques. The breast has real female breast size, skin color and elastic softness. Institutional permission will be requested for the "Simple breast model" in the basic skills laboratory of the Midwifery Department of Hamidiye Faculty of Health Sciences.

INTERVENTIONS:
Other: Scenario-based high-reality hybrid simulation method — Intervention group students will be practiced with the "Lactation Simulator", a high-reality simulator, in the simulation laboratory, accompanied by a scenario.
  Arms: İntervention group (n:40)

SUMMARY:
This research was planned to examine the effects of hybrid simulation-based breastfeeding consultancy training on midwifery students' psychosocial care competence and communication skills. The research population will consist of second-year students studying at Health Sciences University (SBU), Hamidiye Faculty of Health Sciences (HSBF), Department of Midwifery in the spring semester of the 2023-2024 academic year (N: 80). Students participating in the study will be divided into intervention (n: 40) and control (n: 40) groups according to the computer-assisted simple random sampling technique. Control group students will practice on a simple breast model within the scope of classical education. "Descriptive Information Form", "Psychosocial Care Competency Self-Assessment Scale" and "Communication Skills Scale-Adult Form" will be applied to the students participating in the research.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research.
* Being an active student in the second year of the University of Health Sciences, Hamidiye Faculty of Health Sciences, Department of Midwifery.

Exclusion Criteria:

-Being a passive student in the second year of the University of Health Sciences, Hamidiye Faculty of Health Sciences, Department of Midwifery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  In this form, created by the researchers based on the literature, the participants' age, high school they graduated from, previous simulation training, etc. questions are included.
Psychosocial Care Competence Self-Assessment Scale | 10 minutes
  The scale was developed by Karataş and Kelleci in 2020. The four-dimensional scale, which consists of 18 valid and reliable items and is called "symptom identification", "use of information", "intervention" and "diagnosis", is a 5-point Likert type. Item, internal consistency and test-retest analyzes were used for the reliability of the scale and it was determined that the internal consistency coefficient was 0.93 and its sub-dimensions were between 0.80 - 0.93.
Communication Skills Scale-Adult Form | 10 minutes
  The form of the scale used for adults was created by Korkut Owen and Demirbaş-Çelik (2017) by adapting it to the communication skills scale. The scale consists of 25 items and 5 sub-dimensions. The first subscale, consisting of nine items, is called basic skills and self-expression. The second sub-dimension is called paying attention to communication and consists of five items. The third sub-dimension, called willingness to establish relationships, consists of three items. The fourth sub-dimension, called active listening and non-verbal communication, consists of five items. The last sub-dimension, compliance with communication principles, consists of three items. Cronbach's alpha coefficient was calculated for the internal consistency reliability of the scale and the internal consistency coefficient of the scale was found to be .94.

SECONDARY OUTCOMES:
Psychosocial Care Competence Self-Assessment Scale | 10 minutes
  The scale was developed by Karataş and Kelleci in 2020. The four-dimensional scale, which consists of 18 valid and reliable items and is called "symptom identification", "use of information", "intervention" and "diagnosis", is a 5-point Likert type. Item, internal consistency and test-retest analyzes were used for the reliability of the scale and it was determined that the internal consistency coefficient was 0.93 and its sub-dimensions were between 0.80 - 0.93.
Communication Skills Scale-Adult Form | 10 minutes
  The form of the scale used for adults was created by Korkut Owen and Demirbaş-Çelik (2017) by adapting it to the communication skills scale. The scale consists of 25 items and 5 sub-dimensions. The first subscale, consisting of nine items, is called basic skills and self-expression. The second sub-dimension is called paying attention to communication and consists of five items. The third sub-dimension, called willingness to establish relationships, consists of three items. The fourth sub-dimension, called active listening and non-verbal communication, consists of five items. The last sub-dimension, compliance with communication principles, consists of three items. Cronbach's alpha coefficient was calculated for the internal consistency reliability of the scale and the internal consistency coefficient of the scale was found to be .94.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No